CLINICAL TRIAL: NCT01771692
Title: A Study Into the Effects of Different Ligation Techniques on Orthodontic Mandibular Incisor Alignment
Brief Title: A Randomised Clinical Trial: Conventional Ligation vs Figure of 8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rachel Little (Other)
Responsible Party: Sponsor-Investigator, Rachel Little, Specialty Registrar in Orthodontics, University of Birmingham
Organization: University of Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIT001
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Malocclusion
Keywords: Orthodontics
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional ligation (Active Comparator): Modules ligated in a conventional manner (figure of 0)
  Interventions: Other: Extraction; Other: Non extraction
- Figure of 8 ligation (Active Comparator): Modules ligated in a figure of 8 configuration
  Interventions: Other: Extraction; Other: Non extraction

INTERVENTIONS:
Other: Extraction — Extraction of teeth in the lower arch as part of the orthodontic treatment plan
Other: Non extraction — Non extraction in the lower arch as part of the orthodontic treatment plan

SUMMARY:
Fixed braces (appliances) are used to straighten the malalignment of teeth. There has been a lot of research into the factors that can affect the speed of alignment of teeth but there has been very little research on how different techniques of wire attachment to the brace (ligation) can affect this.

The randomised clinical trial of 100 patients aims to compare the speed of alignment of the lower (mandibular) front teeth (incisors) using two different techniques over a period of 12 weeks. Both techniques use the conventional small elastic rings (modules) that are placed over each metal square (bracket) but they will be tied in a different configuration for each group. We will also observe any differences in the distances between the corresponding teeth either side of the lower jaw for each group and the bracket failure rates.

DETAILED DESCRIPTION:
The research protocol has been devised by Rachel Little (Specialty Registrar in Orthodontics), under the supervision of Mr David Spary (Consultant in Orthodontics) and Dr Ashish Dhopatkar (Head of Orthodontics, Birmingham Dental School).

Purpose:

In this study I intend to find out whether friction plays a part in lower incisor alignment by comparing different ligation techniques. If I can show that the speed of alignment is affected by different techniques, this will be an important finding for orthodontic treatment.

Aims:

This study aims to determine whether increased friction caused by ligation with figure of eight modules effects the speed of lower incisor alignment.

Recruitment and consent:

100 orthodontic patients (n=50 per group) who have attended a new patient clinic at Burton Hospital and who require correction for the malalignment of their teeth with a fixed appliances will be selected. Potential participants will be invited to take part in the study and will be given verbal and written information. If they agree to participate, written consent will be obtained. All patients will be competent and capable of making the decision. All patients in this study will be under 16 years of age, and so parental/legal guardian consent will be obtained. The patients will be able to withdraw from the study at any time, should they not wish to continue participating.

Method:

Participants will be randomly allocated to either the conventional module group (figure of O) or the figure of 8 module group, following consent for participation in the trial. Randomisation will use the method of block randomisation. Allocation will be undertaken by a non-clinician.

The plan is to use the study models (replica of the patient's teeth made out of plaster) from the pre treatment records as the baseline data then take an additional mould (impression) of the lower teeth only at each of the participants normal orthodontic appointments at six and twelve weeks after the appliances have been put on.

All measurements required will be taken from these study models using digital callipers, after the impressions have been cast in the laboratory.

Benefits of treatment:

• Improved appearance and function of the teeth

Risks of treatment:

* Tooth decay and gum disease (this can be prevented with good oral hygiene and low sugar intake)
* Discomfort
* Breakages
* Relapse (if retainers are not worn after the fixed appliances are removed)
* Root shortening

Confidentiality:

The study models that will be analysed will be stored in the patient's model box along with their notes in a locked office.

At no point during this research will personal details be disclosed to any persons not directly involved with providing orthodontic care.

Conflict of interest:

No conflict of interest is known or expected to arise during this study.

At the end of the study:

A summary sheet of the findings of this study will be made available to participants on request.

ELIGIBILITY:
Inclusion Criteria:

* Patients at Burton Hospital
* 12-15 years of age at the start of treatment
* No medical contraindications
* Permanent dentition
* Mandibular incisor irregularity of 5-10mm (using Little's irregularity index)
* No other therapeutic intervention e.g. elastics, coils
* Informed consent gained

Exclusion Criteria:

* Presence of a craniofacial syndrome
* Patients already participating in a research study

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Little's irregularity index. | up to12 weeks
  Mandibular incisor irregularity index reduction using Little's irregularity index.

SECONDARY OUTCOMES:
Intercanine width. | 0, 6, 12 weeks
  Changes in intercanine widths between the two groups.

OTHER OUTCOMES:
Intermolar width. | 0, 6, 12 weeks
  Changes in intermolar widths between the two groups.
Bracket failure rate. | 0,6,12 weeks
  Compare orthodontic bracket failure rates between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: David J Spary, BDS LDS FDS DOrth FDS Orth, Study Director — Burton Hospitals Foundation Trust
Locations (1):
- Queen's Hospital, Burton Hospitals NHS Foundation Trust, Burton-on-Trent, Staffordshire, United Kingdom